CLINICAL TRIAL: NCT02758444
Title: Effects of Environmental Enteric Dysfunction (EED) on Zinc (Zn) Absorption and Retention in Young Children: Study 2 - Absorption of Zn From a Multi-micronutrient Powder (MNP)
Brief Title: Effects of EED on Zn Absorption and Retention in Children From a MNP
Acronym: ZEED2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14-2430B
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Environmental Enteric Dysfunction; Zinc Deficiency
Keywords: environmental enteric dysfunction; environmental enteropathy; zinc absorption; Bangladesh; toddlers; zinc isotope

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Micronutrient Powder (MNP) + 15 mg Zn (Active Comparator): 1 sachet of Micronutrient Powder (MNP) + 15 mg Zn will be added to a single meal on study day 8
  Interventions: Dietary Supplement: Micronutrient Powder (MNP) + 15 mg Zn
- MNP + 10 mg Zn (Active Comparator): 1 sachet of MNP + 10 mg Zn will be added to a single meal on study day 8
  Interventions: Dietary Supplement: MNP + 10 mg Zn
- MNP + 5 mg Zn (Active Comparator): 1 sachet of MNP + 5 mg Zn will be added to a single meal on study day 8
  Interventions: Dietary Supplement: MNP + 5 mg Zn
- MNP without Zn (Placebo Comparator): 1 sachet of MNP without Zn will be added to a single meal on study day 8
  Interventions: Dietary Supplement: MNP without Zn

INTERVENTIONS:
Dietary Supplement: Micronutrient Powder (MNP) + 15 mg Zn — Children will have the supplement powder added to one meal on study day 1. Absorption of zinc from this meal will be measured using zinc stable isotope techniques.
  Arms: Micronutrient Powder (MNP) + 15 mg Zn
Dietary Supplement: MNP + 10 mg Zn — Same as above except MNP will contain 10 mg Zn
  Arms: MNP + 10 mg Zn
Dietary Supplement: MNP + 5 mg Zn — Same as above except MNP will contain 5 mg Zn
  Arms: MNP + 5 mg Zn
Dietary Supplement: MNP without Zn — Same as above except MNP will not contain Zn
  Arms: MNP without Zn

SUMMARY:
The overall objective is to determine the impact of EED on total daily zinc absorption of young Bangladeshi children (18-24 months of age) in an austere setting with high rates of diarrhea, stunting, and micro-nutrient deficiencies..

DETAILED DESCRIPTION:
Participating children are screened for EED using the lactulose:mannitol ratio test and assigned to one of two groups: +EED or -EED. After assignment to one of the two groups, proposed subjects will be randomized to one of four supplement groups: Micronutrient powder (MNP) with 15 mg Zn, MNP with 10 mg Zn, MNP with 5 mg Zn, and MNP with 0 mg Zn. Children will receive the supplement once with a meal on Day 8 of the study. Absorption of zinc from the supplement and from other non-supplemented meals will be determined using zinc stable isotope technology.

ELIGIBILITY:
Inclusion Criteria:

* Absence of apparent health problems that would impair ability to consume regular diet, to tolerate zinc supplements, or to comply with demands of metabolic studies
* Length for age Z (LAZ) score between -1.5 to -3.0
* Hg ≥ 8

Exclusion Criteria:

* Outside age range
* Hb < 8
* Chronic illness
* Zinc supplement within past 2 weeks (including for treatment of diarrhea or MNP containing zinc)
* Severe stunting and/or severe acute malnutrition (SAM): LAZ <-3; WHZ <-3 or MUAC < 115 or edema

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Total daily absorbed zinc (TAZ) | 1 day
  Measured during the meal to determine the effects of EED on zinc absorption.

SECONDARY OUTCOMES:
Exchangeable zinc pool (EZP) | 1 day
  Size of exchangeable Zn pool (EZP) measured with zinc isotope methods prior to the meal.
Plasma zinc | 1 day
  Measured prior to the meal.
Alkaline phosphatase | 1 day
  Measured prior to the meal.
Serum retinol | 1 day
  Measured prior to the meal.
Methyl malonic acid | 1 day
  Measured prior to the meal.
Vitamin B12 | 1 day
  Measured prior to the meal.
Serum ferritin | 1 day
  Measured prior to the meal.
Soluble transferrin receptors | 1 day
  Measured prior to the meal.
CRP | 1 day
  Measured prior to the meal.
AGP | 1 day
  Measured prior to the meal.
TNF alpha | 1 day
  Measured prior to the meal.
Serum endocab | 1 day
  Measured prior to the meal.
Neopterin | 1 day
  Measured prior to the meal.
Myeloperoxidase | 1 day
  Measured prior to the meal.
Calprotectin | 1 day
  Measured prior to the meal.
alpha 1 antitrypsin | 1 day
  Measured prior to the meal.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Denver, Aurora, Colorado, United States
- icddr,b (International Centre for Diarrheal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Long JM, Mondal P, Westcott JE, Miller LV, Islam MM, Ahmed M, Mahfuz M, Ahmed T, Krebs NF. Zinc Absorption from Micronutrient Powders Is Low in Bangladeshi Toddlers at Risk of Environmental Enteric Dysfunction and May Increase Dietary Zinc Requirements. J Nutr. 2019 Jan 1;149(1):98-105. doi: 10.1093/jn/nxy245. PMID 30624753